CLINICAL TRIAL: NCT02147795
Title: Safety and Effectiveness of a Patient Blood Management (PBM) Program in Surgical Patients
Brief Title: The German Patient Blood Management Network
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Vifor Pharma (Industry); B. Braun Melsungen AG (Industry); CSL Behring (Industry); Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Professor Kai Zacharowski, M.D., Ph.D., FRCA, Professor Kai Zacharowski, M.D., Ph.D., FRCA, Johann Wolfgang Goethe University Hospital
Other Study IDs: PBM01
Record Dates: First submitted 2014-05-13; First posted 2014-05-28 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Clinical Safety of a PBM Program
Keywords: Patient Blood Management; Red Blood Cell Transfusion Practice; Patient Safety; Anemia; Clinical Outcome; perioperative care
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control cohort: Standard care before implementation (pre-implementation)
- PBM cohort: After implementation of PBM program (post-implementation)

SUMMARY:
* This epidemiological trial will determine whether the implementation of a PBM program is safe and effective in terms of clinical outcome compared to a pre-implementation cohort
* Primary endpoint is a composite outcome comprising in-hospital myocardial infarction, stroke, acute renal failure, death of any cause, pneumonia and sepsis until discharge from hospital in patients before and after implementation of the PBM program.
* Secondary endpoints are the length of stay on the intensive care unit, total hospital stay and the quantitative utilization of allogeneic RBC units, platelet concentrates, other blood products (e.g. fresh frozen (therapeutic) plasma), coagulations factors, and cell saver systems during hospital stay.
* The primary aim is to prove non-inferiority of the intervention (PBM) group when compared with the control group stratified by center.

DETAILED DESCRIPTION:
Background: The transfusion of allogeneic red blood cell units might be associated with increased morbidity and mortality due to infectious, immunological, pulmonary and thromboembolic complications. However, transfusion practice currently varies significantly between hospitals and even between physicians and Patient Blood Management programs have not been implemented nationwide in Germany yet. Patient Blood Management (PBM) concepts aim to identify and optimize patients at risk of allogeneic blood transfusions, to promote blood-sparing techniques and restrictive transfusion practices. A rational use of red blood cell concentrates and safe clinical transfusion practice is mandatory. The purpose of the German PBM network is to evaluate the safety of a standardized, evidence-based Patient Blood management concept.

Study Design and Methods: This epidemiological study is a follow-up of a study that is already being carried out in four German university hospitals. This new prospective, multi-centre trial comprises approximately 20 different hospitals of varying size and levels of patient care. A patient-centred, evidence-based Patient Blood Management program will be enrolled in each of these hospitals reforming the care of adult patients undergoing any type of surgery. This PBM program includes the following three main pillars: 1) preoperative optimization of hemoglobin levels in high-risk patients with anaemia, 2) standardization of transfusion practice and transfusion triggers according to evidence-based guidelines and 3) alternatives to transfusion of allogeneic RBC concentrates and blood-sparing techniques (like routine use of cell saver systems, point-of-care diagnostics, optimized coagulation management, restrictive blood sampling).

ELIGIBILITY:
Inclusion Criteria:

* all surgeries with a general or local anaesthetic
* minimum hospital stay of 24 h
* ≥ 18 years

Exclusion Criteria:

* < 18 years
* ophthalmologic or dermatologic or outpatient surgery
* all non-surgical anesthetic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult surgical patients
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2012-01; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome for and after PBM program | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  composite outcome comprising in-hospital myocardial infarction, stroke, acute renal failure, death of any cause, pneumonia and sepsis until discharge from hospital in patients before and after implementation of the PBM program

SECONDARY OUTCOMES:
Length of stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  length of stay on the intensive care unit, total hospital stay
haemotherapy | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  the quantitative utilization of allogeneic RBC units, platelet concentrates, other blood products (e.g. fresh frozen (therapeutic) plasma), coagulations factors, and any other haemotherapy (including use of cell salvage

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Goethe University Hospital, Frankfurt am Main, Hesse
  - University Hospital Würzburg, Würzburg

REFERENCES:
- [Derived] Meybohm P, Schmitt E, Choorapoikayil S, Hof L, Old O, Muller MM, Geisen C, Seifried E, Baumhove O, de Leeuw van Weenen S, Bayer A, Friederich P, Brautigam B, Friedrich J, Gruenewald M, Elke G, Molter GP, Narita D, Raadts A, Haas C, Schwendner K, Steinbicker AU, Jenke DJ, Thoma J, Weber V, Velten M, Wittmann M, Weigt H, Lange B, Herrmann E, Zacharowski K; German Patient Blood Management Network Collaborators. German Patient Blood Management Network: effectiveness and safety analysis in 1.2 million patients. Br J Anaesth. 2023 Sep;131(3):472-481. doi: 10.1016/j.bja.2023.05.006. Epub 2023 Jun 26. PMID 37380568
- [Derived] Schmitt E, Meybohm P, Neef V, Baumgarten P, Bayer A, Choorapoikayil S, Friederich P, Friedrich J, Geisen C, Guresir E, Grunewald M, Gutjahr M, Helmer P, Herrmann E, Muller M, Narita D, Raadts A, Schwendner K, Seifried E, Stark P, Steinbicker AU, Thoma J, Velten M, Weigt H, Wiesenack C, Wittmann M, Zacharowski K, Piekarski F; German PBM Network Collaborators. Preoperative anaemia and red blood cell transfusion in patients with aneurysmal subarachnoid and intracerebral haemorrhage - a multicentre subanalysis of the German PBM Network Registry. Acta Neurochir (Wien). 2022 Apr;164(4):985-999. doi: 10.1007/s00701-022-05144-7. Epub 2022 Feb 26. PMID 35220460